CLINICAL TRIAL: NCT05810714
Title: Increasing CRC Screening Using Audio and Video Brochures: A Pilot Randomized Controlled Trial
Brief Title: Audio and Video Brochures for Increasing Colorectal Cancer Screening Among Adults Living in Appalachia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Mira Katz, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: OSU-21213; NCI-2022-00144 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R21AG061496 (NIH)
Record Dates: First submitted 2023-03-31; First posted 2023-04-12 (Actual); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm I (FIT, usual care) (Active Comparator): Participants receive the FIT kit and usual care on study.
  Interventions: Other: Best Practice; Other: Fecal Immunochemical Test; Other: Survey Administration
- Arm II (FIT, audio brochure, reminder) (Experimental): Participants receive the FIT kit with an audio brochure, disposable gloves and stool collection device, and scheduled reminder on study.
  Interventions: Other: Fecal Immunochemical Test; Behavioral: Health Education; Other: Scheduled Notification; Other: Survey Administration
- Arm III (FIT, video brochure, reminder) (Experimental): Participants receive the FIT kit with a video brochure, disposable gloves and stool collection device, and scheduled reminder on study.
  Interventions: Other: Fecal Immunochemical Test; Behavioral: Health Education; Other: Scheduled Notification; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Arm I (FIT, usual care)
Other: Fecal Immunochemical Test — Receive FIT kit
  Other Names: FIT; iFOBT; immunoassay fecal occult blood test; immunochemical fecal occult blood test; Immunochemical FOBT; immunologic fecal occult blood test
Behavioral: Health Education — Receive audio brochure
  Arms: Arm II (FIT, audio brochure, reminder)
Behavioral: Health Education — Receive video brochure
  Arms: Arm III (FIT, video brochure, reminder)
Other: Scheduled Notification — Receive scheduled reminder
  Other Names: ScheduledNotification
  Arms: Arm II (FIT, audio brochure, reminder); Arm III (FIT, video brochure, reminder)
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial compares audio brochures and video brochures to usual care for increasing colorectal cancer (CRC) screening among adults living in Appalachia. Adults living in rural Appalachia experience increased rates of CRC, possibly due to the unique barriers to screening this population faces, such as lower socioeconomic status, limited health literacy, and less access to healthcare. The fecal immunochemical test (FIT) is a common CRC screening technique which allows individuals to complete the test at home and mail the kit back. A limitation of the current process for FIT screening outreach is that the instruction materials are heavy in text and not appropriate for individuals with limited health literacy. The audio and video brochures used in this clinical trial are instruction materials that have been specially designed to be appropriate for individuals of all health literacy levels. Providing these audio and video brochures with the FIT kits may increase CRC screening among adults living in Appalachia, compared to usual care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Conduct a pilot study of the two developed mail-based FIT outreach interventions versus (vs.) mailed usual care materials to establish acceptability and obtain preliminary efficacy data on increasing CRC screening.

OUTLINE: Participants are randomized to 1 of 3 arms.

ARM I: Participants receive the FIT kit and usual care on study.

ARM II: Participants receive the FIT kit with an audio brochure, disposable gloves and stool collection device, and scheduled reminder on study.

ARM III: Participants receive the FIT kit with a video brochure, disposable gloves and stool collection device, and scheduled reminder on study.

ELIGIBILITY:
Inclusion Criteria:

* Mid-life men and women (50-64 years old)
* Live in Appalachia
* Had a medical visit in the past two years
* Are at average-risk for CRC (no history of CRC, polyps, inflammatory bowel disease, family history of CRC or hereditary CRC syndromes)
* Are not within CRC screening guidelines (no fecal occult blood test/FIT in the past year; flexible sigmoidoscopy in past five years; colonoscopy in past ten years)

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mira Katz, PhD, MPH, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Katz ML, Shoben AB, Newell S, Hall C, Emerson B, Gray DM 2nd, Chakraborty S, Reiter PL. Video brochures in a mailed fecal immunochemical test outreach program provide cancer screening information in a user-friendly format for rural Appalachian community members. J Rural Health. 2024 Jan;40(1):96-103. doi: 10.1111/jrh.12772. Epub 2023 Jun 9. PMID 37296510

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (FIT, Usual Care) | Arm II (FIT, Audio Brochure, Reminder) | Arm III (FIT, Video Brochure, Reminder)
Started | 20 | 42 | 32
Completed | 20 | 42 | 32
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (FIT, Usual Care) | Arm II (FIT, Audio Brochure, Reminder) | Arm III (FIT, Video Brochure, Reminder) | Total
Number analyzed (Participants) | 20 | 42 | 32 | 94
Age, Continuous [Median (Standard Deviation); unit: years] | 58.3 (4.4) | 57.1 (4.3) | 57.1 (4.2) | 57.1 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 22 | 15 | 47
  Male | 10 | 20 | 17 | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 42 | 32 | 94

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants to Return Fecal Immunochemical Test (FIT)
Description: Will estimate FIT return using proportions for each study group. Both comparisons (each intervention compared to control) will be a two-sample test of proportions (intent-to-treat analysis) using a one-sided alpha of 0.1 due to the preliminary nature of the study.
Time Frame: At 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (FIT, Usual Care) | Arm II (FIT, Audio Brochure, Reminder) | Arm III (FIT, Video Brochure, Reminder)
Number analyzed (Participants) | 20 | 42 | 32
Participants | 3 | 4 | 9

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for up to 60 days.
Arm/Group | Arm I (FIT, Usual Care) | Arm II (FIT, Audio Brochure, Reminder) | Arm III (FIT, Video Brochure, Reminder)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/42 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/42 | 0/32
Other Adverse Events (participants affected / at risk) | 0/20 | 0/42 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/14/NCT05810714/Prot_SAP_000.pdf